CLINICAL TRIAL: NCT04811391
Title: Cohort Study to Measure COVID-19 Vaccine Effectiveness Among Health Workers in Albania
Brief Title: COVID-19 Vaccine Effectiveness in Albanian Health Workers
Acronym: COVEAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Public Health, Albania (Other Government)
Collaborators: World Health Organization (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); Southeast Europe Center for Infectious Diseases Surveillance and Control (Unknown); EPICONCEPT (Unknown)
Responsible Party: Sponsor
Other Study IDs: COV-VE-0001
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: vaccine effectiveness; health care worker; Albania
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Vaccinated participants: Participants who have received 2 doses of the pfizer Covid-19 vaccine or 1 or dose of the Astra Zeneca Covid-19 Vaccine
  Interventions: Biological: COVID-19 vaccine
- Unvaccinated participants: Have not received any doses of any form of COVID-19 vaccine

INTERVENTIONS:
Biological: COVID-19 vaccine — Observation of individuals who receive the COVID-19 vaccine (2 doses of PfizerBioNtech COVID-19 vaccine).
  Groups: Vaccinated participants

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the COVID-19 vaccine in hospital based HWs in Albania. This will answer critical questions about the real-world performance of COVID-19 vaccines in one of the key target groups for vaccination.

DETAILED DESCRIPTION:
This protocol describes a prospective one-year cohort study of hospital-based health workers in Albania to evaluate the effectiveness of COVID-19 vaccine in preventing laboratory-confirmed SARS-CoV-2 infection and COVID -19 disease.

The investigators will measure the effectiveness of COVID-19 vaccines against laboratory-confirmed SARS-CoV-2 infection in both symptomatic and asymptomatic hospital health workers.

SARS-CoV-2 infection will be diagnosed using symptom questionnaires and PCR testing. Additionally, serology testing will be obtained over the course of one year, to identify asymptomatic infections.

ELIGIBILITY:
Inclusion Criteria:

* All Health Workers eligible to receive the COVID-19 vaccination according to the national guidelines of Institute of Public Health.
* Health Workers working at Tirana University Hospital "Mother Theresa", University Hospital "Shefqet Ndroqi", Durres Regional hospital and Fier Regional Hospital.
* Health Workers who have already been vaccinated against COVID-19 as part of the early COVID-19 vaccine rollout can be included, as long as information can be collected about the date and type of the vaccine that was administered. However, priority will be given to enrolling Health Workers who have received their COVID vaccine no more than 4 days prior to the day of enrolment in the study.

Exclusion Criteria:

* Health Workers who are not eligible for COVID-19 vaccination or have a contraindication to vaccination should not participate in the study.
* Health Workers who do not work at Tirana University Hospital "Mother Theresa", University Hospital "Shefqet Ndroqi", Durres Regional hospital and Fier Regional Hospital.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be composed of health workers in the above hospitals, eligible for vaccination, with no contraindication to receive COVID-19 vaccine. Health Workers include all categories of staff working in the hospitals, including clinical and non-clinical/administrative staff and staff with direct patient interaction and those without direct patient interaction.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-05-20 (Estimated)

PRIMARY OUTCOMES:
COVID-19 vaccine effectiveness | 12 months
  Data will be collected using weekly symptom questionnaires, COVID-19 PCR confirmation for any symptomatic participant and quarterly serology assessment for all participants to identify N-protein presents to suggest new infection, rather than vaccine induced antibody response.
COVID-19 PCR confirmation | 12 months
  Data will be collected using weekly symptom questionnaires, COVID-19 PCR confirmation for any symptomatic participant and quarterly serology assessment for all participants to identify N-protein presents to suggest new infection, rather than vaccine induced antibody response.

SECONDARY OUTCOMES:
Vaccine effectiveness by age | 12 months
  The enrollment questionnaire includes age of each participant. Data will be stratified by age at the time of analysis.
Vaccine effectiveness by co-morbidities | 12 months
  The enrollment questionnaire will include specific co-morbidities, including (but not limited to) heart disease, autoimmune disease, chronic liver disease and chronic kidney disease. Data will be stratified by co-morbidity at the time of analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Bino, MD, PHD, Principal Investigator — Institute of Public Health
Locations (3):
- Albania (3):
  - Durres Regional Hospital, Durrës
  - Fier Regional Hospital, Fier
  - Tirana University Hospital " Mother Theresa", Tirana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finci I, Rojas Castro MY, Hasibra I, Sulo J, Fico A, Daja R, Vasili A, Kota M, Preza I, Muhlemann B, Drosten C, Pebody R, Lafond KE, Kissling E, Katz MA, Bino S. Primary Series and Booster Coronavirus Disease 2019 Vaccine Effectiveness in a Cohort of Healthcare Workers in Albania During a BA.1 and BA.2 Variant Period, January-May 2022. Open Forum Infect Dis. 2023 Oct 12;10(10):ofad479. doi: 10.1093/ofid/ofad479. eCollection 2023 Oct. PMID 37885795
- [Derived] Sridhar S, Fico A, Preza I, Hatibi I, Sulo J, Kissling E, Daja R, Ibrahim R, Lemos D, Rubin-Smith J, Schmid A, Vasili A, Valenciano M, Jorgensen P, Pebody R, Lafond KE, Katz MA, Bino S. COVID-19 vaccine effectiveness among healthcare workers in Albania (COVE-AL): protocol for a prospective cohort study and cohort baseline data. BMJ Open. 2022 Mar 23;12(3):e057741. doi: 10.1136/bmjopen-2021-057741. PMID 35321895